CLINICAL TRIAL: NCT00813020
Title: A Randomised, Single Centre, Double-blind, Incomplete Block Trial to Test for Equivalence Between Subcutaneous Injections of the GLP-1 Analogue NN9535 in 1 mg/ml, 3 mg/ml and 10 mg/ml Concentrations in Healthy Male Subject
Brief Title: A Clinical Trial Investigating the Comparison of Three Different Concentrations of NN9535 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-3679; 2008-004990-17 (EudraCT Number)
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: semaglutide
- B (Experimental)
  Interventions: Drug: semaglutide
- C (Experimental)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — Comparison of different formulations of the drug, semaglutide: Formulation 1 administered in equimolar doses
  Arms: A
Drug: semaglutide — Comparison of different formulations of the drug, semaglutide: Formulation 2 administered in equimolar doses
  Arms: B
Drug: semaglutide — Comparison of different formulations of the drug, semaglutide: Formulation 3 administered in equimolar doses
  Other Names: NN9535
  Arms: C

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate whether differences exist between three different concentrations of the drug, NN9535, administered in healthy male subjects in equal doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, based on an assessment of medical history, physical examination and clinical laboratory data at screening, as determined by the Investigator
* Body weight between 80 kg and 110 kg (both inclusive)
* Body Mass Index (BMI) between 18 and 27 kg/m2, both inclusive
* Fasting plasma glucose max 108 mg/dl (6.0 mmol/l)

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products
* Previous participation in this trial (randomisation)
* The receipt of any investigational medicinal product within 3 months prior to this trial
* Subjects who have had a clinically relevant illness within 4 weeks of dosing
* History of or presence of cancer, diabetes, or any clinically relevant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders
* Regular smoking as defined by smoking 1 or more cigarettes or the equivalent amount of tobacco pr day, and unable to refrain from smoking during the entire confinement period

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
AUC0-8 (NN9535), the area under the plasma NN9535 plasma-concentration-time curve in the interval 0-8 after investigational medicinal product administration | a 28 day time period

SECONDARY OUTCOMES:
Cmax of the plasma NN9535 curve | a 28 day time period

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Berlin, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com